CLINICAL TRIAL: NCT02192749
Title: Open, Prospective Trial of Treatment of Autism Spectrum Disorders (ASD) Using Intravenous Infusion of Umbilical Cord Tissue Mesenchymal Stem Cells (UC-MSC)
Brief Title: Allogeneic Umbilical Cord Mesenchymal Stem Cell Therapy for Autism
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Translational Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TBS-UCMSC-ASD001
Record Dates: First submitted 2014-07-12; First posted 2014-07-17 (Estimated); Last update posted 2017-10-13 (Actual); Status verified 2017-10

CONDITIONS: Autism
Keywords: autism; umbilical cord; mesenchymal; stem cells
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Umbilical cord mesenchymal stem cells (Experimental)
  Interventions: Biological: Umbilical cord mesenchymal stem cells

INTERVENTIONS:
Biological: Umbilical cord mesenchymal stem cells

SUMMARY:
Allogeneic (not from the subject) human umbilical cord tissue-derived stem cells administered intravenously (IV) in a series of 4 infusions every 3 months over the course of one year is safe and will induce a therapeutic effect in autism patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female
* Ages 6 to 16
* Diagnostic and Statistical Manual of Mental Disorders (DSM IV) diagnosis of autism confirmed by Autism Diagnostic Observation Schedule (ADOS) and/or Autism Diagnostic Interview-Revised (ADI-R)
* No anticipated changes in treatment for the study duration (e.g., diet, nutrients)
* No additional biomedical treatments started 6 weeks prior to enrollment
* No changes in dietary management for 3 months prior to enrollment
* Ambulatory or require minimum support walking, per parent
* Able to sit still for 5 minutes or longer with a preferred toy item, per parent
* Adequate vision and hearing for the purposes of test administration, per parent
* Adequate arm-hand-finger coordination (i.e., able to point) for learning and cognitive tasks used in outcome measurement, per parent
* Stable and controlled mental disorder
* Under the care of a caregiver willing to participate by attending regularly scheduled appointments and completing the necessary measures
* Normal heavy metals test for lead and mercury levels performed within 30 days of first stem cell infusion
* Must provide name and specialty of specialist who has made Autism Spectrum Disorder (ASD) diagnosis
* Adequate financial means to cover $7,200 (US Dollars) plus travel expenses

Exclusion Criteria:

* Significant prematurity at birth (less than 32 weeks gestation); or birth weight significantly below normal for gestational age (SGA - small for gestational age)
* mental retardation
* seizure disorder
* auto-immune conditions
* history of head trauma and other neurological or medical conditions
* Abnormal heavy metals test for lead and mercury performed within 30 days of first stem cell infusion
* Prior stem cell therapy of any kind

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2014-07; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | 89 weeks

SECONDARY OUTCOMES:
Number of participants with a change in disability as measured by the Autism Treatment Evaluation Checklist (ATEC) | 13 weeks, 25 weeks, 37 weeks, 49 weeks, 89 weeks
Number of participants with a change in disability as measured by the Childhood Autism Rating Scale (CARS) | 13 weeks, 25 weeks, 37 weeks, 49 weeks, 89 weeks
Change from baseline macrophage-derived chemokine (MDC) | 13 weeks, 25 weeks, 37 weeks, 49 weeks, 89 weeks
Change from baseline thymus and activation-regulated chemokine (TARC) | 13 weeks, 25 weeks, 37 weeks, 49 weeks, 89 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Nelson Novarro, MD, Principal Investigator; Jorge Paz-Rodriguez, MD, Principal Investigator — Translational Biosciences / Stem Cell Institute Panama
Locations (1):
- Stem Cell Institute, Panama City, Panama